CLINICAL TRIAL: NCT04417712
Title: Lifetech KONAR-MF™ VSD Occluder Post-Market Clinical Follow-Up Study
Brief Title: Lifetech KONAR MFO Post-Market Clinical Follow-Up Study
Status: Completed | Type: Observational
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: LT/TS/45CE-04-01
Record Dates: First submitted 2020-06-02; First posted 2020-06-05 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Ventricular Septal Defect
Keywords: VSD
MeSH Terms: conditions — Heart Septal Defects, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with ventricular septal defect: All patients who signed informed consent and are implanted with a KONAR-MF™ VSD Occluder device will undergo follow-up (FU) evaluations as per local hospital standards and corresponding IFU which is expected to be at the following time points post-implant:
  * Before discharge
  * 1-3 months after the Procedure
  * 6 months after the procedure
  * 12 months after the procedure
  Interventions: Device: KONAR-MF™ VSD Occluder

INTERVENTIONS:
Device: KONAR-MF™ VSD Occluder — All patients will be implanted with a KONAR-MF™ VSD Occluder in accordance with the instructions for use (IFU).

SUMMARY:
The purpose of the study is to collect real-world data on patient outcomes and evaluate the procedural success and performance of the Lifetech KONAR-MF™ VSD Occluder for patients with ventricular septal defect (VSD).

DETAILED DESCRIPTION:
This is a non-randomized prospective post-marketing clinical follow-up study (PMCFS) in order to evaluate the feasibility and safety of the Lifetech KONAR-MF™ VSD Occluder device used for patients with ventricular septal defect. The implantation should be performed in accordance with the instructions for use (IFU).

ELIGIBILITY:
Inclusion Criteria:

1. Patients have a clinically relevant ventricular septum defect (VSD) by Echocardiography and/or X-ray examination according to current clinical standards and center-specific protocols.
2. The patient should be older than 6 months of age and a bodyweight heavier than 8kg.
3. Defect diameter (by 2D Echocardiography): The size of the VSD is larger than or equal to 2mm and less than 10mm.
4. Upper margin of VSD to aortic valve distance >2 mm for models 6-4, 8-6, 10-8, 12-10, 14-12 and >2.5mm for models 5-3, 7-5, 9-7, in case of PmVSD.
5. Only left to right shunt of the ventricular shunt.

Exclusion Criteria:

1. Any contraindication mentioned in the corresponding IFU*.

   * Note: In IFU, contraindications for The KONAR-MFTM VSD Occluder are as follows:

     1. Patient has extensive congenital cardinal anomaly which can only be adequately repaired by cardiac surgery.
     2. Presence of thrombus at the intended site of implant, or documented evidence of venous thrombus in the vessels through which access to the defect is gained.
     3. Active endocarditis or other infections-producing bacteria.
     4. The implant of KONAR-MFTM VSD Occluder would cause an obvious interference with the aortic valve or the atrioventricular valve.
     5. Patients with severely increased pulmonary vascular resistance and a right-to-left shunt and patients with documented irreversible pulmonary vascular disease.
     6. Patients with contraindications to anti-platelet therapy or agents.
2. The patient does present with an aortic valve prolapsing into the VSD.
3. Currently participating in other investigational drugs- or device studies.
4. The patient who is pregnant, planning to become pregnant, or breastfeeding.
5. Patients don't give informed written consent for the procedure.
6. Patient with other cardiac anomalies by surgery therapy.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ventricular septal defect (VSD).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Accurate success rate | From implant attempt to 12-month post-procedure.
  VSD closure without complication (dislocation, hemolysis, AVB, device-related valve dysfunction, thrombosis, infection, or endocarditis) and no or only mild residual shunt after 12 months of follow-up.
Procedure successful | From implant attempt to 12-month post-procedure.
  The optimal position of the VSD with appropriate closure rate at echocardiographic examination. No or only tiny or without residual shunt and absence of device-related aortic or atrioventricular valve reflux.

SECONDARY OUTCOMES:
Rate of device and procedure-related serious adverse events (SAE). | From implant attempt to 12-month post-procedure.
  Rate of device and procedure-related serious adverse events (SAE) during 12 months post-procedure.
Rate of complete atrioventricular block (cAVB) or any arrhythmia needed for pacemaker implantation, device removal, or any kind of medical treatment. | From implant attempt to 12-month post-procedure.
  Rate of complete atrioventricular block (cAVB) or any arrhythmia needed for pacemaker implantation, device removal, or any kind of medical treatment in patients within 12 months post-implantation.
Rate of incomplete closure at the 12-month follow-up. | At 12-month follow-up.
  Rate of incomplete closure at the 12-month follow-up: significant shunt will be defined as ≥ moderate or indicating treatment (surgical or interventional). The residual shunt will be defined by color Doppler echocardiography and will measure the shunt size according to prior published classification.
Rate of device deficiencies. | From implant attempt to 12-month post-procedure.
  Rate of device deficiencies (including device malfunction, failures, and non-conformances) during 12 months post-procedure.
Incidence within 12 months post-implantation | From implant attempt to 12-month post-procedure.
  Incidence within 12 months post-implantation for:
  1. Hemolysis including any drop in hemoglobin (Hb) of >2.5 g/dl within 24 hours and Severe acute hemolysis, which is defined as Hb ≤5 g/dl or received blood transfusion according to the clinical judgment of the study physician.
     Hemolysis can be excluded by sample urine within 24 hours post-implantation. If hemolysis might be suspected, blood sampling (blood count incl. hemoglobin) should be initiated according to SOP or clinical practice.
  2. Thromboembolism: thrombosis of device or vascular access that requires thrombolytic therapy;
  3. Migration of the occlude requiring device removal;
  4. Embolization of the occluder requiring device removal.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Schubert, Principal Investigator — Heart- and Diabetescenter NRW
Locations (4):
- Germany (3):
  - 103 - Herz- und Diabeteszentrum NRW / Heart and Diabetes Center NRW, Bad Oeynhausen
  - 101 - Deutsches Herzzentrum der Charité/ German Heart Institute Berlin, Berlin
  - 102 - Deutsches Herzzentrum München/ German Heartcenter Munich, Munich
- IRCCS Policlinico San Donato, Milan, Italy